CLINICAL TRIAL: NCT01793376
Title: Development of Niv Score of Capsule Endoscopy in Patients With Crohn's (CECDAIic)
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-208-1
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis This study is designed as an integral part of the development of a new CE score for Crohn's disease.

The SB (small bowel) CD (Crohn's Disease)Niv score (CECDAI) is an established and validated CD score for SB involvement. In order to expand this score to the colon, this study will aim to develop the colonic score and later on will be combined with the already established SB score in order to achieve a full CE gut score for Crohn's disease Proposed Design This is a retrospective study in which up to 30 videos of colon Crohn's disease subjects who have undergone the Colon 2 CE procedure will be evaluated.

These cases will have evidence of large and / or small bowel Crohn's disease The chosen videos will be marked for CD lesions by the site The de-identified marked videos will be scored by 4 independent experienced endoscopists, blinded to the results of the standard workup procedures, according to the colonic and CECDAIic new scores

ELIGIBILITY:
Inclusion Criteria:

* videos of colon Crohn's disease subjects who have undergone the Colon 2 CE procedure will be included.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: videos of colon Crohn's disease subjects who have undergone the Colon 2 CE procedure will be included.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The inter-observer variability of the new CD Colonic Score, between four reviewers in Crohn's Disease patients with large bowel involvement | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yaron Niv, Prof., Principal Investigator — Rabin MC